CLINICAL TRIAL: NCT06408714
Title: Comparison of Nalmefene Hydrochloride Injection and Naloxone Hydrochloride Injection for the Treatment of Recurrent Respiratory Depression After Suspected Acute Opioid Overdose in the Emergency Department
Brief Title: Nalmefene vs Naloxone for the Treatment of Recurrent Respiratory Depression After Opioid Overdose
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Caitlin Bonney, Assistant Professor of Emergency Medicine, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNM24-157
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Opioid Overdose; Opiate Overdose
Keywords: opioid overdose; opiate overdose; drug overdose; naloxone; nalmefene; respiratory depression
MeSH Terms: conditions — Opiate Overdose; Drug Overdose; Respiratory Insufficiency | interventions — nalmefene; Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nalmefene (Experimental): Nalmefene Rescue Study Arm Treatment:
  Subjects will receive study drug if they exhibit respiratory depression (defined as respiratory rate less than 8 breaths per minute and/or end-tidal carbon dioxide measurement of greater than 50 mm Hg) lasting for longer than 10 seconds. Respiratory support with bag-valve mask and/or supplemental oxygen will be provided while the study drug is being prepared. Nalmefene will be administered as per intervention description.
  Interventions: Drug: Nalmefene Injection
- Naloxone (Active Comparator): Naloxone Rescue Arm Treatment:
  Subjects will receive study drug if they exhibit respiratory depression (defined as respiratory rate less than 8 breaths per minute and/or end-tidal carbon dioxide measurement of greater than 50 mm Hg) lasting for longer than 10 seconds. Respiratory support with bag-valve mask and/or supplemental oxygen will be provided while the study drug is being prepared. Naloxone will be administered as per intervention description.
  Interventions: Drug: Naloxone Injection

INTERVENTIONS:
Drug: Nalmefene Injection — Subjects in this arm will be administered intravenous nalmefene with a dosing scheme of:
  0.5 mg Nalmefene IV
  If an adequate response (increase in RR of at least 5 breaths per minute and minimum respiratory rate of 12 breaths per minute or reduction in ETCO2 to 40 mm Hg) is not attained after 2 minutes, an additional 1.0 mg nalmefene will be administered.
  If an adequate response is not attained after an additional 2 minutes of observation, naloxone may be administered as a rescue agent at the treating physician's discretion.
  Other Names: Nalmefene; Nalmefene hydrochloride; Nalmefene HCl
  Arms: Nalmefene
Drug: Naloxone Injection — Subjects in this arm will be administered intravenous naloxone with a dosing scheme of:
  0.4 mg Naloxone IV
  If an adequate response (increase in RR of at least 5 breaths per minute and minimum respiratory rate of 12 breaths per minute or reduction in ETCO2 to 40 mm Hg) is not attained after 2 minutes, an additional 0.4 mg of naloxone will be administered.
  If an adequate response is not attained after an additional 2 minutes of observation, naloxone may be administered as a rescue agent at the treating physician's discretion.
  Other Names: Naloxone; Naloxone HCl; Naloxone hydrochloride
  Arms: Naloxone

SUMMARY:
The goal of this clinical trial is to compare naloxone to nalmefene for the treatment of opioid overdose in adults. The main questions it aims to answer are:

* Does nalmefene lower the number of doses of medicine participants need to treat opioid overdose?
* When participants are given nalmefene instead of naloxone, do they have fewer complications of opioid overdose such as being admitted to the hospital or having a breathing tube inserted?

Researchers will compare nalmefene to naloxone for the treatment of opioid overdose. Nalmefene and naloxone are both approved medicines to treat opioid overdose.

Participants who are brought to the emergency department after an opioid overdose will be given a dose of either nalmefene or naloxone if their breathing slows down again after an opioid overdose. Participants will:

* Stay in the emergency department for 8 hours after receiving a dose of nalmefene or naloxone.
* Receive a phone call 7 days after their emergency department to check on how they are doing.

Background information:

Naloxone (also known as Narcan) and nalmefene are opioid blocking medicines. When someone overdoses on an opioid, such as heroin or fentanyl, their breathing slows down or stops and they can die. By giving naloxone or nalmefene, the effect of the opioid can be blocked and the person can start breathing again. Naloxone is the most commonly used medicine to reverse an opioid overdose. The effect of naloxone lasts about an hour, and patients may need more than one dose of naloxone to keep them breathing. Sometimes patients overdose, get a dose of naloxone and wake up, and then some time later their breathing slows down again and they need another dose of naloxone. This can happen because the effect of the opioid they took lasts longer than the effect of the naloxone.

The effect of nalmefene lasts longer than naloxone, about four hours. If a person gets nalmefene, their opioid may wear off before the nalmefene wears off and they might not need any more doses of a reversal medicine. Both naloxone and nalmefene are approved medicines for treating opioid overdose.

Often, when a person overdoses on an opioid, someone gives them naloxone right away and then they are brought to the emergency department. In the emergency department, they are watched for several hours to make sure they don't stop breathing again when their naloxone wears off. If they do stop breathing again, they are given another dose of naloxone. In this study, participants will be given either nalmefene or naloxone if their breathing slows down while they are in the emergency department.

DETAILED DESCRIPTION:
1. Study Design This is an open-label prospective randomized single center study comparing nalmefene to naloxone in the treatment of recurrent respiratory depression from opioids.
2. Number of Subjects

   We will enroll 37 patients in the nalmefene group and 37 patients in the naloxone group, for a total of 74 patients.

   Based upon our feasibility study of naloxone administrations in the ED, 344 patients received naloxone in the ED during a two-year period (2021-2022), corresponding to approximately 14 patients per month. (Note that this is likely their 2nd dose of naloxone, as nearly all patients arrive via EMS and we presume received naloxone by EMS.) We estimate that 75% of patients who receive opioid antagonist treatment during EMS transport or shortly after ED arrival will be capable of providing informed consent in the ED. We estimate that up to 50% may decline to participate. Based on these parameters, we estimate enrolling 5.4 patients per month or 96 subjects over the 18 month enrollment period.

   In our power and sample size analysis we estimated we would need to enroll 62 subjects. We added a 20% increase in our sample size to account for subjects that might not stay for the observation period, for a total of 74 patients.

   To enroll 74 patients, we will screen 220 patients for eligibility and consent.

   Sample size justification:

   We conducted power analyses with varying scenarios for a noninferiority clinical trial comparing nalmefene versus naloxone. For a redosing rate (p1) of 0.33 for naloxone and a redosing rate (p2) of 0.05 for nalmefene, a significance level (alpha) of 0.025, and a margin of noninferiority of -0.02, we would need 31 patients in each, respectively. This would give us a total of 62 patients to achieve a power of 0.8. We will enroll 20% extra patients, or 37 patients in each group, in anticipation of patients not completing the observation period or the study, for a total of 74 patients.
3. Study Timelines

   * The duration of an individual subject's participation in the research: 7 days
   * Initial visit: emergency department visit with observation of 8 hours after emergency department arrival or until discharge, whichever comes first.
   * Second evaluation: phone follow up at 7 days
   * The duration anticipated to enroll all subjects: 1.5 years

8. Research Setting Study site: Single center study at the University of New Mexico Hospital Adult Emergency Department. UNMH is the only academic medical center, Level I trauma center, and stroke center in New Mexico. UNMH is also the safety net hospital for the greater Albuquerque area. The UNMH ED saw over 102,000 patients in 2022, of whom ~58,000 were seen in the adult ED.

Biological samples will be processed by TriCore Laboratories, the contracted laboratory service for UNM HSC. Xylazine and nitazene testing will be performed at NMS Labs (nmslabs.com).

9. Resources Available

The UNMH emergency department is staffed 24 hours a day with licensed emergency physicians ("attending physicians"). Attending physicians will be responsible for medical decision-making and ordering and evaluation of necessary diagnostics and therapeutics for study participants.

Resources:

The Department of Emergency Medicine maintains a workforce of full-time trained research staff specializing in research subject identification and recruitment. All staff are trained in human subject research, good clinical practices and Basic Science Laboratory level 1 and 2 (BSL 1-2) procedures. Staff are able to accommodate regular night and weekend coverage to ensure adequate staffing to respond to potential subject enrollments.

All study personnel are required to maintain current human subject protections and good clinical practices certifications and complete and document study specific training and delegation on study training and delegation logs.

Pharmacy Resources: The UNMH investigational drug service is used in this study. The investigational drug service allows for the secure storage and dispensation of investigational drugs in accordance with applicable state and federal regulations and institutional policies.

Laboratory resources: The UNM HSC Clinical and Translational Sciences Center (CTSC) contract laboratory will be used for the processing and storage of research samples. The CTSC contract laboratory provides secure 24-hour access to calibrated continuous temperature monitored freezers, centrifuge and BSL-2 lab bench space. Quanititative Nalmefene and Xylazine testing will be performed by NMS labs.

12. Study Procedures

* Screening: Study subjects will be recruited from the University of New Mexico Hospital Emergency Department. Research Assistants (RAs) will identify patients seen in the ED by reviewing the electronic medical record (EMR) tracking board, notification by secure messaging system of arriving patients, and by provider referral.
* Informed Consent: Patients who are determined to meet all inclusion and none of the exclusion criteria will be approached about informed consent by a trained IRB-approved study team member. For additional detail on informed consent see Section 21 Consent Process.
* Enrollment and Randomization: Patients who provide written informed consent are considered enrolled in the study. Subjects will be asked to complete demographics, medical history and prior and concomitant medications by survey at the time of enrollment. Blood Alcohol Content (BAC) will be measured by Breathalyzer. Participants will then be randomized using the UNM Health Sciences REDCap randomization tool to either nalmefene or standard care (naloxone) treatment arms. Research staff will be blinded to randomization.
* Blood Collection: Blood collection for serum testing for co-ingestants, xylazine, and nitazenes will be performed after enrollment. Blood collection for research testing will involve no more than 15 mL (1 tablespoon) in up to 3 tubes at one timepoint.
* Subject Follow-Up: RAs will remain present with the patient in the peri-dosing period to observe and record any adverse events, including any occurrence of precipitated withdrawal or recrudescence, for no less than 8 hours after emergency department arrival or until emergency department discharge, whichever comes first. Subjects will be contacted by phone 7 days (+/- 2 days) after enrollment to assess for recurrence of opioid overdose symptoms, repeat emergency department visits or hospitalizations and occurrence of adverse events.
* Data Acquisition: Demographics, medical history and prior and concomitant medications, adverse events will be collected by subject interview/survey and/or observation in the ED. All other data elements such as details related to medication, laboratory and imagining results, diagnosis and information on subsequent discharge and/or hospitalization or return visit to the emergency department will be captured from the subjects EMR.

  13. Data Analysis Plan We will use an intention-to-treat analysis. For the primary outcome, we will compare the proportion of subjects experiencing the primary endpoint (respiratory depression requiring opioid antagonist treatment) using the Newcombe's method for the difference between two proportions1, adjusted for a non-inferiority framework as the initial analysis.

As we expect that the time to event (respiratory depression) will differ between the two treatment arms, we will also compare the risk of recurrent respiratory depression using a failure time analysis. Failure time analysis (also known as survival analysis) allows us to assess the risk of a failure event (here, recurrent respiratory depression) while adjusting for observations that are time dependent and of varying length. Failure time analyses also correctly account for incomplete observations because of a study ending or loss of subjects to follow-up (we anticipate that some subjects may not stay for the full observation period). For the initial analysis, we anticipate using nonparametric techniques, such as Kaplan-Meier curve estimation and log-rank tests to assess for differences in recurrent respiratory depression between the two arms. Most frequently, failure time analysis is used in situations where only one event occurs (such as a diagnostic endpoint, disease cure, or death) and the subject then is withdrawn from the study. In the proposed study, subjects can experience multiple failure events (recurrent episodes of respiratory depression) because a rescue therapy (naloxone or nalmefene) is available. After completing the initial non-parametric analyses, we propose an additional analysis that will allow us to take advantage of the likelihood that subjects may have more than one endpoint. Since multiple events can occur within the same subject, calculation of standard errors and statistical inference need to account for the correlation between observations in the same individual. The method we propose using does this precisely and we have used this method for a different poisoning/antidote study.2,3 With this method, the point estimate of the relative risk is not affected by the correlation between repeat measurements within the same individual, and therefore can be calculated using a proportional hazards model. All analyses will use the R statistical language.

14. Provisions to Monitor the Data to Ensure the Safety of Subjects Data monitor services will be provided by the University of New Mexico Hospitals Clinical Trials Operations Office and supervised by Leslie Byatt, BA, CCRC, PCP. The study data monitor is not directly affiliated with the study.

Safety monitoring will be provided by Snehal Bhatt, MD. Dr Bhatt is an experienced addiction medicine physician. Dr Bhatt is affiliated with the University of New Mexico School of Medicine.

All study subjects will be asked to stay in the UNMH Emergency Department for the duration of the 8 hour observation period. All adverse events will be recorded for the duration of the 8 hour observation period. All adverse event information will be prepared in summary, deidentified, and provided to the safety monitor on the following schedule for review:

Review 1: After completion of the 3rd subject enrollment (4% of subjects enrolled) Review 2: After completion of the 10th subject enrollment (14% of subjects enrolled) Review 3: After completion of the 26th subject enrollment (35% of subjects enrolled) Review 4: After completion of the 42nd subject enrollment (57% of subjects enrolled) Review 5: After completion of the 74th and final subject enrollment (100% of subjects enrolled) This safety monitor review schedule is subject to change in the event that the safety monitor raises concerns that merit more frequent reviews.

All serious adverse events will be gathered through the day 7 follow-up. In the event of a serious adverse event (SAE) that is determined to be unexpected and possibly or probably related to the investigational product, enrollment will be temporarily stopped until the safety monitor has reviewed and provided recommendations related to ongoing study conduct. Once any recommendations, if any, have been addressed, the study may continue. Initial SAE reports have to be reported within 24 hours of the identification of an SAE, follow-up attempts will be made as needed within 3 days or no later than 14 days from the initial report, if additional information becomes available this will be processed as per our procedures. . All SAE's will be followed to resolution. All SAE information will be gathered in a detailed summary report and transmitted to the safety monitor for review. Only SAEs will be forwarded to Drug Safety mailbox at AEreport2@pharma.com. The investigator will be using the following definitions for AEs, SAEs and reportable new information. The SAE report from will include start and stop date, whether or not it was unexpected, concise identification according to the Common Terminology for the Categorization of Adverse Events (CTCAE), detailed narrative description including why it is determine to meet the SAE definition below, any medical interventions to address the SAE, the events relationship to the study intervention, and report type (initial, follow-up or final). All SAE's must be reviewed by the principal investigator prior to submission to the safety monitor for review.

Adverse Event (AE): Any untoward or unfavorable medical occurrence in a human study participant, including any abnormal sign (e.g. abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participants' involvement in the research, whether or not considered related to participation in the research.

Serious Adverse Event (SAE): Any adverse event that:

* Results in death
* Is life threatening, or places the participant at immediate risk of death from the event as it occurred
* Requires or prolongs hospitalization
* Causes persistent or significant disability or incapacity
* Results in congenital anomalies or birth defects
* Is another condition which investigators judge to represent significant hazards

A pregnancy is not by definition an SAE but is handled as an SAE because it is not a condition that should occur during the clinical trial, requires the subject to be discontinued from the study, and requires ongoing monitoring of the pregnancy by the PI. Abnormal pregnancy outcomes are considered as reportable SAEs. SAEs associated with pregnancy outcome include, but are not limited to:

* Pregnancy losses (e.g., spontaneous abortion, late fetal death, elective termination)
* Life-threatening developments (e.g., placental abruption, fetal distress) • Congenital anomalies
* Neonatal fatality, any event resulting in maternal hospitalization /prolonged hospitalization or maternal fatality.

Any female subject who becomes pregnant while participating will be withdrawn from the study but will be contacted to determine the pregnancy outcome.

The study team will promptly report all unanticipated problems that meet the following criteria to the UNM HSC HRRC within 5 business days of identification as reportable information. Defined by DHHS 45 CFR part 46 as any incident, experience, or outcome that meets all of the following criteria:

* unexpected, in terms of nature, severity, or frequency, given (a) the research procedures that are described in the protocol-related documents, such as the IRB-approved research protocol and informed consent document; and (b) the characteristics of the study population;
* related or possibly related to participation in the research (in this guidance document, possibly related means there is a reasonable possibility that the incident, experience, or outcome may have been caused by the procedures involved in the research);
* suggests that the research places participants or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

Subjects in the trial will receive clinical care in the UNM Hospital Emergency Department. As subjects are also patients being treated for the effects of opioid intoxication, all will receive standard of care. Standard care includes: establishing intravenous access to provide additional medication to reverse respiratory depression, end-tidal carbon dioxide monitoring, pulse oximetry, electrocardiographic monitoring, and vital sign monitoring. All subjects will receive care from the ED treatment team. The ED team consists of a board-certified EM faculty member, resident physicians, advanced practice providers, emergency medicine pharmacists, and registered nurses. All subjects in the trial will be treated in appropriate clinical spaces within the ED. A full spectrum of standard emergency equipment is readily available (e.g., airway adjuncts, advanced monitoring, etc.

15. Withdrawal of Subjects The study medical clinician must apply their clinical judgement to determine if an adverse event is of sufficient severity to require that the participant be withdrawn from further study participation. The study medical clinician should consult with the site Principal Investigator, the Co-Investigator, and/or Medical Monitor as needed. If necessary, a study medical clinician may suspend any trial treatments and institute the necessary medical therapy to protect a participant from any immediate danger.

A participant may also voluntarily withdraw from treatment due to what they perceive as an intolerable adverse event or for any other reason. If a voluntary withdrawal is requested, the participant will be asked to complete an end-of-medication visit to assure safety and to document end-of-medication outcomes and will be given recommendations for medical care and/or referrals to treatment as necessary.

A participant may withdraw from any portion of the protocol (e.g. serum collection for expanded toxicology testing) but complete other aspects of the study.

A participant may withdraw from the study at any time.

16. Data Management/Confidentiality All study data will be stored in accordance with all applicable state and federal regulations and in accordance with institutional requirements. All subject source information will be stored N:\Research-Studies network drive.

The research team will have access to the patient's medical record to abstract elements from the patient's chart relevant to the study, including patient disposition and additional AE and SAE's and 7 day follow-up data.

Zip codes will not be recorded. Information abstracted as part of the research study will not include direct patient identifiers (i.e., name, MRN, FIN, address). Subjects will be identified by a unique study number. A link between the patient's identifying information will remain secured and stored apart from study data on the N: drive. This data will include substance abuse information.

Data from this study will not be publicly available.

All study data will be entered into UNM Health Sciences REDcap, a secure web application for building and managing online surveys and databases. After study closure all data will be stored in the N:\Research-studies network drive.

All study specimens will be labeled with a unique study ID only and stored only for the duration of testing described in this protocol. Specimens will not be banked for this study and will only be accessible to IRB approved members of the study team.

No data will be collected by audio or video recording. Data will not include photographs. This study is not funded by the NIH. Data will be retained for a period of 6 years from the date the study is complete and then destroyed. No minors will be included in this study.

17. Data and Specimen Banking Neither data nor specimens will be banked for this study.

18. Risks to Subjects

Study related risks include medication risks, study procedures risks and loss of confidentiality.

Medication risks associated with the use of naloxone and nalmefene are very similar and may include precipitation of severe opioid withdrawal, recurrent respiratory and central nervous system depression, nausea, vomiting, fever, dizziness, headache, chills, and vasodilation (relaxing/dilation of blood vessels). Other risks associated with reversal of opioid overdose include cardiac related risks such as pulmonary edema (fluid in the lungs), cardiovascular instability, hypotension (low blood pressure, hypertension (high blood pressure), tachycardia (fast heart rate), ventricular fibrillation (irregular heart beat). Risks associated with the use of nalmefene and naloxone in pregnant people include precipitated withdrawal in the fetus.

Risks associated with study procedures, which include a study blood draw are minimal. They include pain, bruising, infection, lightheadedness, fainting, blood clots, and bleeding or other discomforts at the draw site.

Risks associated with the possible loss of confidentiality may include emotional discomfort or stress.

19. Potential Benefits to Subjects There are no known benefits to subjects.

20. Recruitment Methods Potential subjects will be identified for participation in the study after presentation to the UNM ED for suspected acute opioid overdose. Based upon our feasibility analyses, we expect that most subjects will arrive via EMS. Our dispatch team uses a secure text messaging system (TigerConnect, https://tigerconnect.com/) to alert designated staff members of pending patient arrivals based off EMS radio reports. These messages typically provide a very brief description of the patient and their condition. A typical message might say: "32 M with RR 4 and sat 80%, now RR 16 and 95% after Narcan. ETA 10 minutes". These messages give the research team the opportunity to proactively identify potential subjects. We currently use a cadre of trained research assistants to monitor our ED tracking board and EMS message alerts, and to provide just-in-time reminders to clinical staff about current studies. We will use these research assistants to aid in subject identification. These RAs are typically able to consent subjects for most studies. Due to the acuity of the event and our current crowded ED state, nearly all patients with an opioid OD requiring active management (supplemental oxygen, BVM, naloxone administration) are moved to our resuscitation area for rapid assessment and stabilization. Once stabilized, patients can be relocated to other spaces in the ED.

Potential subjects will be identified by

* Notification of the study team by a treating physician when a potentially eligible patient presents to the emergency department.
* Research assistants will monitor patient arrival alerts in TigerConnect for potentially eligible patients.
* Research assistants will monitor the UNMH ED tracking board for potentially eligible patients.

  21. Provisions to Protect the Privacy Interests of Subjects Potential subjects will be recruited from the UNM ED. Whenever possible, subjects will be approached in a private setting. The IRB-approved study personnel responsible for approaching the potential subject about informed consent will be responsible for confirming with the patient that they are willing to discuss study participation prior to attempting to obtain informed consent. All study data will be gathered directly from the subject or the subject's chart in a standard patient care area within the UNMH ED or by phone for the 7 day follow-up. If the potential patient expresses privacy concerns before or during participation, it will be the IRB-approved research team member's responsibility to address that concern to the best of their ability and to document any steps taken to address these concerns on a study notes page. Study personnel may have limited ability to address privacy concerns in certain circumstances and if they are unable to address the potential subject's privacy concerns the potential subject will be excluded from participation.

  22. Economic Burden to Subjects Subjects will be responsible for all costs associated with standard care they receive as part of the emergency department visit. The research will cover all costs associated with research procedures. UNM will not charge study subjects, insurers or any other third parties for any study activities covered by the protocol and paid for by Purdue Pharma. Purdue Pharma shall not be responsible for the care or treatment of any illness or injury occurring to any study subject regardless of whether such costs are otherwise covered by such study subject's medical or hospital insurance, government program or other third party payor.

  24. Compensation for Research-Related Injury Research related injury is not expected in this study. We do not expect to see higher rates of research related injury in the nalmefene or naloxone treatment arms, as such there are not funds set aside for compensation in the event of research related injury. In the event of research related injury subjects are responsible for seeking care. UNM Hospital will provide care in the event of research related injury but subjects may seek or request care elsewhere. Subjects will be responsible for the cost of that care. Purdue Pharma shall not be responsible for the care or treatment of any illness or injury occurring to any Study subject regardless of whether such costs are otherwise covered by such Study subject's medical or hospital insurance, government program or other third party payor.

  25. Consent Process Subjects are considered enrolled once they have signed and dated the IRB-approved informed consent form. The consent process will take place in patient care areas in the UNMH ED. Details related to maintaining patients' privacy are described in Section 21. Provision to Protect the Privacy Interests of Subjects. Consent will be obtained by IRB-approved study team members who are trained and delegated this task on study training and delegation logs. The IRB-approved study team member obtaining informed consent will be responsible for documenting their consent discussion with the potential participant on a study notes page and confirm the subject's ability to give informed consent by completing the UCSD Brief Assessment of Capacity to Consent (attached). Only English-speaking subjects will be enrolled in the study. Spanish-only speaking subjects will not be enrolled because it is rare for patients in the population being studied to only speak Spanish.The study will not permit consent by a legally authorized representative and will not be enrolling those who are cognitively impaired or unable to give consent. This study will not include minors under the age of 18 years.

  26. Documentation of Consent Subject consent will be documented on a hard copy informed consent form. Details of the circumstances of informed consent will be recorded on a study notes page. Information substantiating a subject's ability to give informed consent will be recorded on a UCSD Brief Assessment of Capacity to Consent for each subject at the time of consent.

  27. Study Test Results/Incidental Findings Individual subject research specific information will not be shared with subjects. Any information relevant to their medical care will be provided by their care team. The study will not generate any incidental findings that are relevant to the subjects' care.

  28. Sharing Study Progress or Results with Subjects We do not intend to provide subjects with a summary of the trial progress while the study remains underway. We do not intend to provide subjects with a summary of the study results after the study is complete.

  29. Inclusion of Vulnerable Populations As this study involves subjects who have experienced a suspected opioid overdose, it is likely that the sample will be enriched with subjects who are economically or educationally disadvantaged. The informed consent form is specifically composed to minimize use of complicated language to the greatest degree possible. IRB approved study team members obtaining informed consent are responsible for ensuring the voluntariness of participation by reiterating the voluntariness of participation, confirming subject understanding and eliciting questions during the process of informed consent.

  33. Drugs or Devices The UNMH investigational drug service is used in this study. The investigational drug service allows for the secure storage and dispensation of investigational drugs in accordance with applicable state and federal regulations and institutional policies. The drugs used in this investigation will be used on-label. The investigational drug service will also ensure that the subjects are not billed for the investigational product.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years) presenting to the UNM ED after a suspected acute opioid overdose event requiring at least one dose of naloxone.

Exclusion Criteria:

* age <18 years
* non-English speaking
* unable to or unwilling to provide consent to research participation
* allergy to naloxone
* allergy to nalmefene
* inability to establish IV access
* prior enrollment in the current study
* no working phone number for follow-up contact
* buprenorphine administration during the ED visit prior to enrollment.
* known pregnancy at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Recurrent respiratory depression | Within 8 hours of intervention
  Recurrent respiratory depression requiring repeat treatment with an opioid antagonist. Respiratory depression is defined as a respiratory rate (RR) <8 breaths per minute or end-tidal CO2 (ETCO2)> 50 mm Hg.

SECONDARY OUTCOMES:
Precipitated withdrawal | Within 8 hours of intervention
  • Proportion of subjects experiencing precipitated withdrawal (Clinical Opioid Withdrawal Scale greater than 5 within 20 minutes) after treatment with an opioid antagonist. The Clinical Opioid Withdrawal Scale, or COWS, ranges from 0 to 48, with a higher score signifying worse withdrawal.
Serious adverse event | Within 8 hours of intervention
  • Proportion of subjects experiencing a serious adverse event (likely admission to the hospital, typically for pulmonary edema, methadone overdose, or co-ingestions requiring extended observation).

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Bonney, MD, Principal Investigator — University of New Mexico Health Sciences Center
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Newcombe RG. Interval estimation for the difference between independent proportions: comparison of eleven methods. Stat Med. 1998 Apr 30;17(8):873-90. doi: 10.1002/(sici)1097-0258(19980430)17:83.0.co;2-i. PMID 9595617
- [Background] Wei LJ, Lin DY, Weissfeld L. Regression analysis of multivariate incomplete failure time data by modeling marginal distributions. J Am Stat Assoc. 1989;84:1065-1073.
- [Background] McLaughlin SA, Crandall CS, McKinney PE. Octreotide: an antidote for sulfonylurea-induced hypoglycemia. Ann Emerg Med. 2000 Aug;36(2):133-138. doi: 10.1067/mem.2000.108183. PMID 10918104